CLINICAL TRIAL: NCT00667485
Title: A Phase I Study of Rapamycin (Sirolimus) With Bevacizumab in Patients With Advanced Malignancies
Brief Title: Rapamycin Plus Bevacizumab in Advanced Cancers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15878B; AVF4180s
Record Dates: First submitted 2008-04-24; First posted 2008-04-28 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Advanced Cancer; Metastatic Cancer
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Sirolimus; Fluid Therapy; Bevacizumab; Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Weekly Rapamcyin (Experimental): Rapamycin (liquid) taken weekly and Bevacizumab (IV infusion ) once every 3 weeks
  Interventions: Drug: Rapamycin (liquid); Drug: Bevacizumab
- Daily Rapamycin (Experimental): Daily oral rapamycin (tablets) and Bevacizumab (IV infusion)once every 3 weeks
  Interventions: Drug: Bevacizumab; Drug: Rapamycin (Tablets)

INTERVENTIONS:
Drug: Rapamycin (liquid) — Weekly Rapamycin (liquid) 90mg (dose will be split 45mg on Day 1 and Day 2 of each week)
  Other Names: sirolimus; Rapamune
  Arms: Weekly Rapamcyin
Drug: Bevacizumab — Multiple doses (dose depends on time of study entry) given by IV once every 3 weeks
  Other Names: Avastin
Drug: Rapamycin (Tablets) — Daily oral rapamycin (tablets) - 2 doses will be tested 4mg and 6mg
  Other Names: sirolimus; Rapamune
  Arms: Daily Rapamycin

SUMMARY:
The goal of this trial is to determine the toxicity and maximum dose of rapamycin and bevacizumab given together to subjects with advanced cancers. This study will also look at the pharmacokinetics and antitumor activity of the combination.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic or unresectable solid tumor for which standard treatments do not exist or are no longer effective
* Performance status of 0-1
* Measurable or non-measurable disease
* Life expectancy of at least 12 weeks
* No anticipated need of other cancer treatments within the next 4 weeks
* 18 years or older
* Negative pregnancy test for women able to have children, agreement to use a medically accepted birth control method while receiving the study drugs and for at least 2 weeks after stopping, not breast feeding
* Ability to understand and willingness to sign a written informed consent document
* No evidence of bleeding diathesis
* Patients without lung cancer receiving anti-coagulation treatment can participate
* Adequate organ and marrow function:

  * ALT and AST less than or equal to 2.5 times the institutional ULN (less than 5 times for patients with liver involvement)
  * hemoglobin at least 9g/dL
  * absolute neutrophil count at least 1,500/µL
  * platelets at least 100,000/µL
  * total bilirubin less than or equal to 1.5 times the institutional ULN
  * creatinine less than or equal to 1.5 times the institutional ULN

Exclusion Criteria:

* Prior treatment with both bevacizumab and an mTOR inhibitor is not allowed. Prior treatment with both bevacizumab OR mTOR inhibitor (including rapamycin) is allowed. Patients who had a grade 3 or greater side effect with either bevacizumab or an mTOR inhibitor cannot take part in this study.
* Chemotherapy or Immunotherapy within the 4 weeks of study start
* Radiotherapy within 14 days of study start
* Cannot be receiving any other investigational drugs or any other cancer treatments while on study (with the exception of androgen ablating agents for patients with prostate cancer).
* Patients with squamous non-small cell lung cancer (NSCLC)
* Patients with lung cancer or lung metastases:

  * on full dose anticoagulation
  * taking 325mg aspirin per day
  * on non-steroidal anti-inflammatory agents
* HIV positive patients receiving combination anti-retroviral therapy are excluded due to potential for serious infections while taking marrow suppressing agents
* Ongoing illness or medical exclusions, including but not limited to:

  * active or ongoing infection
  * symptomatic congestive heart failure
  * uncontrolled hypertension despite optimal medical management
  * cardiac arrhythmia except paroxysmal atrial fibrillation
  * psychiatric illness/social situations that would limit compliance with study requirements
  * history of organ allograft, bone marrow or peripheral blood stem cell transplant
  * known or suspect allergy to bevacizumab or rapamycin
  * seizure disorder treated with steroid or anticonvulsant therapy
  * thrombotic or embolic events within 6 months of starting study
  * pulmonary hemorrhage/bleeding within 12 weeks of starting study (grade 3 event within 4 weeks of first dose of drug). Patients with a history of pulmonary hemorrhage/bleeding cannot be on full dose anticoagulation.
  * pulmonary fibrosis or interstitial lung disease
  * serious non-healing wound, ulcer or bone fracture
  * Major surgery, open biopsy or a traumatic injury within 4 weeks of starting study drug
  * anticipated need for major surgery while on-study
  * current use of any herbal supplements or rifampin (rifampicin)
  * prior history of hypertensive crisis or hypertensive encephalopathy
  * history of myocardial infarction or unstable angina within 6 months of starting study
  * known CNS disease
  * significant vascular disease
  * symptomatic peripheral vascular disease
  * evidence of bleeding diathesis or coagulopathy
  * core biopsy or other minor surgical procedure (except placement of vascular access device) within 7 days of starting study
  * history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months of study start
  * proteinuria at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2008-04; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Toxicity | 3 weeks

SECONDARY OUTCOMES:
Response | 6 weeks
Pharmacokinetics | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ezra Cohen, MD, Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States